CLINICAL TRIAL: NCT02590523
Title: Intracameral Antibiotic Safety Study
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of antibiotic availability
Sponsor: Panhandle Eye Group, LLP (Other)
Responsible Party: Principal Investigator, Sloan W. Rush, MD, Physician, Panhandle Eye Group, LLP
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Intracameral Antibiotics; Cataract Surgery; Phacoemulsification; Endophthalmitis; Vancomycin; Moxifloxacin
MeSH Terms: conditions — Endophthalmitis | interventions — Vancomycin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- A: Vancomycin (Experimental): Intracameral vancomycin injection given at conclusion of cataract case
  Interventions: Drug: Vancomycin
- B: Moxifloxacin (Experimental): Intracameral moxifloxacin injection given at conclusion of cataract case
  Interventions: Drug: Moxifloxacin
- C: Placebo (Placebo Comparator): Intracameral placebo injection with BSS given at conclusion of cataract case
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vancomycin — Intracameral vancomycin injection during cataract surgery
  Arms: A: Vancomycin
Drug: Moxifloxacin — Intracameral moxifloxacin injection during cataract surgery
  Arms: B: Moxifloxacin
Drug: Placebo — Intracameral placebo injection with BSS during cataract surgery
  Arms: C: Placebo

SUMMARY:
The goal of this study is to determine the safety (but not efficacy in preventing infection) of sterile-packaged and pre-loaded injectable solutions of both vancomycin and moxifloxacin at certain dosages and concentrations as prepared by a compounding pharmacy when used intracamerally at the time of cataract surgery.

DETAILED DESCRIPTION:
Use of injectable prophylactic intracameral antibiotics during cataract surgery is gaining popularity worldwide due to the growing body of scientific evidence supporting its use. To date, there is no sterile-packaged antibiotic that has FDA approval for this indication. Surgeons using intracameral injectable antibiotics during cataract surgery must use existing pharmaceuticals off-label and/or rely on imprecise and sub-sterile compounding pharmacies to dispense these types of medications. Both of these scenarios may pose significant risk to patient safety.

Description of the Treatment: Approximately 0.2 mL of either pre-loaded sterile vancomycin hydrochloride 1% solution (1 mg/0.1 mL of normal saline) or moxifloxacin hydrochloride 0.15% solution (150 μg/0.1 mL of normal saline) is injected into the eye with a blunt tip 30 gauge cannula through a small clear corneal incision as the last step in the cataract removal procedure. The purpose of the treatment is for prophylaxis against post-operative infections and endophthalmitis.

Description of Effector Pharmaceuticals/Drugs: Vancomycin is a hydrophilic glycopeptide antibiotic that has been well studied in many different forms: intravenous injectable, oral tablet and even topical eye drop solutions. It is derived from Actinobacteria spp. Moxifloxacin is a synthetic fourth generation fluoroquinolone and has, likewise, been available in many forms including intravenous injectable, oral tablet and topical eye drop solutions. In this study, a contracted compounding pharmacy will produce the two pharmaceutical agents at the concentration/dosage mentioned above under the USP 797 guidelines.

Therapeutic Mode of Action: The primary mode of action for vancomycin is inhibition of cell wall synthesis in gram positive bacteria. The molecule forms hydrogen bonds with terminal amnio acid moieties of the N-acetylmuramic acid (NAM) and N-acetylglucosamine (NAG) polymer. The disruption to the polymerization and cross-linking of NAM-NAG complexes undermines the structural integrity of the bacterial organism leading to bacteriostasis and eventually cell death. The primary mode of action for moxifloxacin is inhibiting DNA gyrases, both type II topoisomerase and topoisomerase IV. These enzymes are essential for bacterial DNA replication to occur.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of visually significant cataract
* Appropriate candidate for cataract surgery

Exclusion Criteria:

* Not willing to undergo an investigational treatment or are unable to cooperate well enough to safely perform the procedure under the protocol guidelines
* Has known allergies to the pre-/intra-/post-operative medications or preservatives in the medications will also be excluded
* Has significant ocular co-morbidities in one or both eyes which may include (but is not limited to): advanced glaucoma, advanced or active macular degeneration, Fuchs corneal dystrophy, prior corneal transplantation, advanced diabetic eye disease, history of retinal detachment or any patient that would require billing a complex cataract procedure for any reason
* Has a known history of a condition which causes an immuno-compromised host state

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse event | 3 months

SECONDARY OUTCOMES:
Postoperative visual acuity measured by best spectacle corrected | 3 months
  best spectacle corrected

OTHER OUTCOMES:
Endothelial cell count measured by specular microscopy | 3 months
  specular microscopy
Rate of postoperative complication | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rush Eye, Amarillo, Texas, United States